CLINICAL TRIAL: NCT03507205
Title: Korean Nationwide Multicenter Pooled Registry of Drug-Eluting Stents
Acronym: Grand-DES
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Investigator, Seoul National University Hospital
Other Study IDs: Grand-DES
Record Dates: First submitted 2018-04-15; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
Keywords: Everolimus; Sirolimus; Zotarolimus; Biolimus; Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- HOST-BIOLIMUS-Korea-3000: Active prospective registration of patients receiving biodegradable polymer-coated biolimus-eluting stents (BP-BES; Biomatrix, Biomatrix Flex, Nobori)
  Interventions: Device: Biomatrix; Biomatrix Flex; Nobori
- EXCELLENT-PRIME: Active prospective registration of patients receiving durable polymer-coated everolimus-eluting stents (DP-EES; Xience Prime)
  Interventions: Device: Xience Prime
- EXCELLENT Prospective cohort: Active prospective registration of patients receiving durable polymer-coated everolimus-eluting stents and sirolimus-eluting stents (Xience V/Promus; Cypher)
  Interventions: Device: Xience V/Promus; Cypher
- HOST-RESOLINTE: Active prospective registration of patients receiving durable polymer-coated zotarolimus-eluting stents (DP-ZES-RI; Resolute Integrity)
  Interventions: Device: DP-ZES-RI
- RESOLUTE-Korea: Active prospective registration of patients receiving durable polymer-coated zotarolimus-eluting stents (DP-ZES; Endeavor; Resolute)
  Interventions: Device: Endeavor; Resolute

INTERVENTIONS:
Device: Biomatrix; Biomatrix Flex; Nobori — Biodegradable polymer-coated biolimus-eluting stents
  Other Names: BP-BES
  Groups: HOST-BIOLIMUS-Korea-3000
Device: Xience Prime — Durable polymer-coated everolimus-eluting stents
  Other Names: DP-EES-Prime
  Groups: EXCELLENT-PRIME
Device: Xience V/Promus; Cypher — Durable polymer-coated everolimus-eluting stents; Sirolimus-eluting stents
  Other Names: DP-EES; SES
  Groups: EXCELLENT Prospective cohort
Device: DP-ZES-RI — Durable polymer-coated zotarolimus-eluting stents
  Other Names: Resolute Integrity
  Groups: HOST-RESOLINTE
Device: Endeavor; Resolute — Durable polymer-coated zotarolimus-eluting stents
  Other Names: DP-ZES
  Groups: RESOLUTE-Korea

SUMMARY:
The objective of this study is to evaluate the long-term efficacy and safety of coronary stenting with the various types of drug-eluting stents (DES) and to determine clinical device and procedural success during commercial use of DES in the real world.

The investigators will compare EES (Xience V/Promus and Xience Prime), SES (Cypher), ZES (Resolute Integrity, Endeavor Resolute, Endeavor), and BES (Biomatrix, Biomatrix Flex, and Nobori).

DETAILED DESCRIPTION:
The Grand Drug-Eluting Stent (Grand-DES) Registry incorporated five different multicenter registries in South Korea. The EXCELLENT prospective cohort and the EXCELLENT-PRIME registry were dedicated for durable polymer-coated everolimus-eluting stents (DP-EES; Xience V/Promus and Xience Prime) or 1st-generation sirolimus-eluting stents (Cypher), the HOST-RESOLINTE and RESOLUTE-Korea registry for durable polymer-coated zotarolimus-eluting stents (DP-ZES; Resolute Integrity and Endeavor Resolute) or 1st-generation Endeavor-ZES, and the HOST-BIOLIMUS-3000-Korea registry for biodegradable polymer-coated biolimus-eluting stents (BP-BES; Biomatrix, Biomatrix Flex, and Nobori). During the period of 2008 through 2014, all registries enrolled all-comers without any exclusion criteria except patient's withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* The patient agrees to participate in this study by signing the informed consent form.
* Alternatively, a legally authorized patient representative may agree to the patient's participation in this study and sign the informed consent form.

Exclusion Criteria:

* There are no exclusion criteria for this registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 17,286 patients derived from a population of patients receiving percutaneous coronary intervention for ischemic heart disease will be enrolled in the present registry.
Sampling Method: Non-Probability Sample
Enrollment: 17286 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | 36 months
  A composite of cardiac death, target-vessel myocardial infarction, and clinically-driven target lesion revascularization

SECONDARY OUTCOMES:
Patient-oriented composite outcome | 36 months
  A composite of all-cause death, all-cause myocardial infarction, and any repeat revascularization
All-cause death | 36 months
  All-cause death
Cardiac death | 36 months
  Cardiac death
All-cause myocardial infarction | 36 months
  All-cause myocardial infarction
Target-vessel myocardial infarction | 36 months
  Target-vessel myocardial infarction
Any repeat revascularization | 36 months
  Any repeat revascularization
Clinically-driven target vessel revascularization | 36 months
  Clinically-driven target vessel revascularization
Clinically-driven target lesion revascularization | 36 months
  Clinically-driven target lesion revascularization
Definite or probable stent thrombosis | 36 months
  Definite or probable stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (37):
- South Korea (37):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Sejong General Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Hallym University Sacred Heart Hospital, Anyang
  - Kosin University Gospel Hospital, Busan
  - Dankook University Hospital, Cheonan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Gwangju Christian Hospital, Gwangju
  - Kwangju Veterans Hospital, Gwangju
  - Chonbuk National University Hospital, Iksan
  - Wonkwang University Hospital, Iksan
  - Inje University Ilsan Paik Hospital, Ilsan
  - National Health Insurance Corporation Ilsan Hospital, Ilsan
  - Inha University Hospital, Inchon
  - Chungbuk National University Hospital, Jeonju
  - Presbyterian Medical Center, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Bundang CHA Medical Center, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Ewha Womans University Medical Center Mokdong Hospital, Seoul
  - Gangbuk Samsung Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Boramae Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Yonsei University Medical Center, Seoul
  - St. Carollo Hospital, Suncheon
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park J, Han JK, Kang J, Chae IH, Lee SY, Choi YJ, Rhew JY, Rha SW, Shin ES, Woo SI, Lee HC, Chun KJ, Kim D, Jeong JO, Bae JW, Yang HM, Park KW, Kang HJ, Koo BK, Kim HS. The Clinical Impact of beta-Blocker Therapy on Patients With Chronic Coronary Artery Disease After Percutaneous Coronary Intervention. Korean Circ J. 2022 Jul;52(7):544-555. doi: 10.4070/kcj.2021.0395. Epub 2022 Apr 4. PMID 35491482
- [Derived] Hwang D, Park J, Yang HM, Yang S, Kang J, Han JK, Park KW, Kang HJ, Koo BK, Kim HS. Angiographic complete revascularization versus incomplete revascularization in patients with diabetes mellitus. Cardiovasc Diabetol. 2022 Apr 19;21(1):56. doi: 10.1186/s12933-022-01488-7. PMID 35439958
- [Derived] Kim M, Park KW, Lee HS, Ki YJ, Kang J, Kim CH, Han JK, Yang HM, Kang HJ, Koo BK, Kim HS. The validation of the dual antiplatelet therapy score in East Asians receiving percutaneous coronary intervention with exclusively second generation drug-eluting stents. Catheter Cardiovasc Interv. 2021 Sep;98(3):E332-E341. doi: 10.1002/ccd.29682. Epub 2021 Apr 5. PMID 33817960
- [Derived] Kang J, Park KW, Lee HS, Zheng C, Rhee TM, Ki YJ, Chang M, Han JK, Yang HM, Kang HJ, Koo BK, Kim HS. Relative Impact of Clinical Risk Versus Procedural Risk on Clinical Outcomes After Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2021 Feb;14(2):e009642. doi: 10.1161/CIRCINTERVENTIONS.120.009642. Epub 2021 Feb 5. PMID 33541106
- [Derived] Zheng C, Kang J, Yang HM, Han JK, Park KW, Kang HJ, Koo BK, Kim HS. Safety and Efficacy of Glycoprotein IIb/IIIa Inhibitors in Patients With Acute Myocardial Infarction in the Presence of Intracoronary Thrombus: An Analysis From the Grand Drug-eluting Stent Registry. Clin Ther. 2020 May;42(5):954-958.e6. doi: 10.1016/j.clinthera.2020.02.022. Epub 2020 Mar 26. PMID 32224030